CLINICAL TRIAL: NCT05291312
Title: Comparison of Endoscope-Assisted Coblation Adenoidectomy to Conventional Curettage Adenoidectomy in Terms of Postoperative Evaluation of Middle Ear Pressure
Brief Title: EACA VS CCA in Postoperative Evaluation of Middle Ear Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MMRafaat, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: EACA AND CCA
Record Dates: First submitted 2022-03-01; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Adenoid Hypertrophy
MeSH Terms: interventions — Adenoidectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endoscopic assisted coblation (Other)
  Interventions: Procedure: Adenoidectomy with endoscopic assisted coblation (EACA) and Adenoidectomy with conventional curettage (CCA)
- conventional curettage (Other)
  Interventions: Procedure: Adenoidectomy with endoscopic assisted coblation (EACA) and Adenoidectomy with conventional curettage (CCA)

INTERVENTIONS:
Procedure: Adenoidectomy with endoscopic assisted coblation (EACA) and Adenoidectomy with conventional curettage (CCA) — IN the (EACA) group slight head flexion position will be given to the patients and Boyle-Davis retractor will be placed to keep the mouth open. The soft palate will be elevated upward by inserting a plastic feeding catheter.. IN the (CCA) group, by orotracheal intubation , Boyle-Davis mouth retractor will be used to provide mouth opening

SUMMARY:
Is to evaluate the effect on Eustachian Tube (ET) and changes in middle ear pressure in early period after adenoidectomy by using Endoscopic Assisted Coblation Adenoidectomy (EACA) VS Conventional Curettage Adenoidectomy (CCA)

DETAILED DESCRIPTION:
Adenoid hypertrophy is a common condition in children causing symptoms such as mouth breathing, nasal discharge, snoring, sleep apnea, and hypo nasal speech. It also plays a role in the pathogenesis of rhinosinusitis, recurrent otitis media, and otitis media with effusion. Currently, adenoidectomy is one of the most commonly performed pediatric surgical procedures worldwide. Although there is still poor evidence in the literature, recurrent upper respiratory infections, otitis media with effusion, and obstructive sleep apnea syndrome are considered to be the main indications of adenoidectomy . Conventional curettage adenoidectomy (CCA) is a widely adopted method for over a hundred years. Conventional curettage adenoidectomy is performed blindly via adenoid curette; this may be associated with residual adenoid tissue existence and increased postoperative morbidity including, Eustachian tube dysfunction, inadvertent injury to peripheral tissue and postoperative bleeding . An ideal adenoidectomy technique should be safe, quick, easy, and provide decreased postoperative complication and morbidity .Recently Adenoidectomy can be carried out with several techniques such as electrocautery, bipolar coagulation, radiofrequency ablation, and coblation techniques .

Eustachian tube dis function (ETD) can develop due to surgical trauma , edema in surrounding tissues and clots in early period following adenoidectomy surgery performed with curettage technique .

ELIGIBILITY:
Inclusion Criteria:

- Pediatric patients presented with adenoid hypertrophy who undergoing primary adenoidectomy with or without tonsillectomy , with the following criteria:

* Age: between ( 5-14 years )
* With or without chronic tonsillitis
* Clinicaly Normal tympanic membrane without secretory otitis media .

Exclusion Criteria:

* Patients with the following criteria will be excluded from the study :
* Patients with secretory otitis media .
* Previous adenoidectomy.
* Previous ear surgery, cleft palate, Down's syndrome, congenital malformation of the ear and cholesteatoma.
* Recurrent upper respiratory tract infection.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
compare Endoscopic Assisted Coblation Adenoidectomy to Conventional Curettage Adenoidectomy in Terms of Postoperative Evaluation of Middle Ear Pressure . | one month
  To compare and analyze changes in middle ear pressure in early period after Adenoidectomy by using Endoscopic assisted Coblation Adenoidectomy to Conventional Curettage Adenoidectomy by using tympanogram

REFERENCES:
- [Result] Turkoglu Babakurban S, Aydin E. Adenoidectomy: current approaches and review of the literature. Kulak Burun Bogaz Ihtis Derg. 2016 May-Jun;26(3):181-90. doi: 10.5606/kbbihtisas.2016.32815. PMID 27107607
- [Result] Thornval A. Wilhelm Meyer and the adenoids. Arch Otolaryngol. 1969 Sep;90(3):383-6. doi: 10.1001/archotol.1969.00770030385023. No abstract available. PMID 4896109
- [Result] Atilla MH, Kaytez SK, Kesici GG, Bastimur S, Tuncer S. Comparison between curettage adenoidectomy and endoscopic-assisted microdebrider adenoidectomy in terms of Eustachian tube dysfunction. Braz J Otorhinolaryngol. 2020 Jan-Feb;86(1):38-43. doi: 10.1016/j.bjorl.2018.08.004. Epub 2018 Sep 25. PMID 30322828
- [Result] Caylakli F, Hizal E, Yilmaz I, Yilmazer C. Correlation between adenoid-nasopharynx ratio and endoscopic examination of adenoid hypertrophy: a blind, prospective clinical study. Int J Pediatr Otorhinolaryngol. 2009 Nov;73(11):1532-5. doi: 10.1016/j.ijporl.2009.07.018. Epub 2009 Sep 3. PMID 19732970
- [Result] Bidaye R, Vaid N, Desarda K. Comparative analysis of conventional cold curettage versus endoscopic assisted coblation adenoidectomy. J Laryngol Otol. 2019 Apr;133(4):294-299. doi: 10.1017/S0022215119000227. Epub 2019 Mar 19. PMID 30885281
- [Result] Elnashar I, El-Anwar MW, Basha WM, AlShawadfy M. Objective assessment of endoscopy assisted adenoidectomy. Int J Pediatr Otorhinolaryngol. 2014 Aug;78(8):1239-42. doi: 10.1016/j.ijporl.2014.04.031. Epub 2014 May 14. PMID 24930960
- [Result] Juneja R, Meher R, Raj A, Rathore P, Wadhwa V, Arora N. Endoscopic assisted powered adenoidectomy versus conventional adenoidectomy - a randomised controlled trial. J Laryngol Otol. 2019 Apr;133(4):289-293. doi: 10.1017/S0022215119000550. PMID 31046870
- [Result] Clemens J, McMurray JS, Willging JP. Electrocautery versus curette adenoidectomy: comparison of postoperative results. Int J Pediatr Otorhinolaryngol. 1998 Mar 1;43(2):115-22. doi: 10.1016/s0165-5876(97)00159-6. PMID 9578120